CLINICAL TRIAL: NCT03841188
Title: Calcium Intake Improvement After Nutritional Intervention in Pediatric Patients With Osteogenesis Imperfecta
Brief Title: Nutritional Interventional in Pediatric Patients With Osteogenesis Imperfecta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-0585
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Osteogenesis Imperfecta
Keywords: osteogenesis imperfecta; Nutritional intervention; calcium intake
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Orientation (Other): The patients received a nutritional orientation with emphasis in food rich in calcium
  Interventions: Other: Nutritional orientation

INTERVENTIONS:
Other: Nutritional orientation — Nutritional orientation with emphasis in rich calcium food

SUMMARY:
BACKGROUND: In several bone disorders, adequate calcium intake is a coadjuvant intervention to regular treatment. Osteogenesis imperfecta (OI) is a collagen disorder with a range of symptoms, ranging from fractures to minimum trauma, and is typically treated with bisphosphonates. This study aims evaluate the impact of a nutritional intervention (NI) on dietary calcium intake, bone mineral density (BMD)in pediatric patients with OI. METHODS: Interventional cohort study was designed with a NI. Dietary calcium intake, anthropometry and clinical feature was assessed at baseline including anthropometry, basal metabolic rate (BMR), BMD, Food guidance form was developed and sent to patients by mail. After 12 months, patients' clinical features were reassessed and compared with baseline data. RESULTS: Fifty-two children and adolescents were enrolled. A significant increase in total calcium intake (g), the percentage of adequate calcium intake (%), number of cups of milk ingested, were observed after NI. Was detected a positive correlation between the variation of BMD and milk consumption in patients treated with bisphosphonate. CONCLUSION: Was observed an increase in calcium intake in patients with OI. This finding demonstrates the importance of nutrition therapy as part of a multidisciplinary treatment approach for bone health.

DETAILED DESCRIPTION:
Nutrition Intervention NI was performed at three nutritional visits (baseline, 6 and 12 months). Clinical features were evaluated at baseline, including anthropometric measurements, basal metabolic rate (BMR), BMD An indirect calorimetry test was performed to estimate the BMR of each participant. Dietary intake was assessed using daily food intake report completed by participants on three non-consecutive days. The frequency of consumption and amount of calcium intake were evaluated using a food frequency questionaire (FFQ) with emphasis on foods rich in calcium. Based on these data, the nutritional needs for each subject were calculated, and personalized food guidance (including recipes rich in calcium) was delivered by mail.

In the second visit, at 6 months after baseline, adaptations were made to food guidance according to the needs of each patient, doubts about feeding were clarified and the importance of a diet rich in calcium was reinforced.

On the third visit, at 12 months after baseline, dietary calcium intake, anthropometric measurements, , BMD were re-evaluated.

Calcium Intake Calcium intake was assessed using an FFQ adapted to calcium intake applied before and after the NI. In the present study, the focus was on the consumption of foods high in calcium, such as milk, yogurt, and cheese. To establish the percentage of the adequacy of intake, the values obtained from the FFQ were compared with the Estimated Average Requirement (EAD) and Recommended Dietary Allowances (RDA).

The FFQ for calcium intake was composed of milk (1 cup = 175 ml), 1 yogurt (120 ml), and cheese (1 medium slice = 30 g). These foods were classified according to the consumer (as D, daily; W, weekly, and M, monthly) and indicating the number of times (1 to 10) and the size of the corresponding portion, if greater, equal or less than the given portion (according to a poster with color photos to illustrate the portion size of each food source of calcium).

Consumption of glasses of milk and soda were also evaluated according to quantity and frequency (For milk, 0 = does not consume, 1 = consume < 1 cup per day, 2 = consume 1 to 2 cups/day, and 3 = consume 3 or more cups of milk/day; for soda, 1 = consume daily, 2 = consume only on weekends or 2 times/week, 3 = consumes less than 1 day/week, and 4 = does not consume).

Clinical Data Clinical data were obtained during the enrollment and included age, gender, OI type, use of bisphosphonates, and calcium intake.

Anthropometric Data and Basal Metabolic Rate Anthropometric measurements (weight and height) were measured and evaluated according to the z-score proposed by the World Health Organization WHO. The length was measured in the supine position in children smaller than 1 m and children could not remain in the standing position. Patients over 1.04 m and unable to remain standing were measured in the supine position. BMI was calculated according to the WHO. The BMR was evaluated through indirect calorimetry and the data was published previously.

Bone Mineral Density BMD was determined before and after the intervention using Dual Energy X-Ray Absorptiometry (DEXA) on a Lunar DXA (GE Healthcare, San Francisco, USA). Bone mineral content (BMC) (g), lumbar spine BMD (L1-L4), and total body BMC (TB) were calculated and expressed as z-scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients from zero to 19 years of patients seen at hospital.
* Diagnosed with osteogenesis imperfecta

Exclusion Criteria:

- Diagnosed with bone disorder

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02-08 (Actual); Primary Completion 2013-05-20 (Actual); Study Completion 2014-02-10 (Actual)

PRIMARY OUTCOMES:
Calcium intake | 12 months
  Was assessed using an food frequency questionaire adapted to calcium intake

SECONDARY OUTCOMES:
Consumption of glasses of milk | 12 months
  Evaluated according to quantity and frequency (For milk, 0 = does not consume, 1 = consume < 1 cup per day, 2 = consume 1 to 2 cups/day, and 3 = consume 3 or more cups of milk/day
Body mass index | 12 months
  Calculation divides an children's weight in kilograms by their height in metres squared.Evaluated according to the z-score proposed by the WHO (2006, 2007)
Bone Mineral Density | 12 months
  Bone mineral density was assessed thought Dual-energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Elza D Mello, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided